CLINICAL TRIAL: NCT02858297
Title: Glucosamine as a Novel Adjunctive Therapy in Oral Lichen Planus: A Pilot, Randomized, Clinical and Immunohistochemical Trial
Brief Title: Glucosamine as a Novel Adjunctive Therapy in Oral Lichen Planus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ola Mohamed Ezzatt, Lecturer of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-RECD 1214403
Record Dates: First submitted 2016-07-26; First posted 2016-08-08 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Oral Lichen Planus
Keywords: Oral lichen planus; Glucosamine; IL-8
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Glucosamine; Triamcinolone Acetonide; Triamcinolone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Glucosamine/Corticosteroid 4 (Experimental): Topical steroid (triamcinolone acetonide 0.1 %) four times per day and (glucosamine sulfate 500 mg) orally three times per day for 8 weeks
  Interventions: Drug: Glucosamine sulfate; Drug: triamcinolone acetonide
- Glucosamine/Corticosteroid 2 (Experimental): Topical steroid (triamcinolone acetonide 0.1 %) twice per day and (glucosamine sulfate 500 mg) orally three times per day for 8 weeks
  Interventions: Drug: Glucosamine sulfate; Drug: triamcinolone acetonide
- Corticosteroid (Active Comparator): Topical steroid (triamcinolone acetonide 0.1 %) four times per day for 8 weeks
  Interventions: Drug: triamcinolone acetonide

INTERVENTIONS:
Drug: Glucosamine sulfate — Glucosamine (GlcN) is an N-deacetyl amino sugar derived from the complete hydrolysis of chitosan with recently reported immunoregulatory capacity and anti-inflammatory effect
  Arms: Glucosamine/Corticosteroid 2; Glucosamine/Corticosteroid 4
Drug: triamcinolone acetonide — Topical corticosteroid
  Other Names: Kenalog in orabase

SUMMARY:
Glucosamine (GlcN) is an N-deacetyl amino sugar derived from the complete hydrolysis of chitosan with recently reported immunoregulatory capacity and anti-inflammatory effect and was administrated orally in osteoarthritis and atopic dermatitis therapy. Given the Oral lichen planus (OLP) T-cell-mediated pathogenesis; this drug seems to be a promising therapeutic option. The investigators compared clinical effectiveness of Glucosamine combined with two topical corticosteroid regimens to that of topical corticosteroid alone in symptomatic OLP and investigated therapeutic mechanism by examining treatment effect on expression of inhibitor kappa kinase alpha (IKKα) and interleukin-8 (IL-8) in OLP lesions.

DETAILED DESCRIPTION:
Thirty patients with Erosive or Atrophic OLP were randomly assigned into Three equal groups to receive combination of topical steroid (triamcinolone acetonide 0.1 %) four times per day and (glucosamine sulfate 500 mg) orally three times per day for 8 weeks (Group I), combination of topical steroid twice daily and glucosamine sulfate 500 mg orally three times per day for 8 weeks (Group II), or topical steroid alone four times per day for 8 weeks (Group III) all patients were followed up for another treatment free 4 weeks observational period. Photographs of the most severe lesion were taken (Marker lesion) in each patient and analyzed for Total Ulcerative Area (TUA), Total Atrophic Area (TAA), and Total Reticular Area (TRA), patients were also assessed using clinical scores (CS) and visual analogue scale (VAS). Pre-treatment and post-treatment specimens were immunohistochemically stained to detect expression of IKKα and IL-8.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and Histologically proven painful Bullous/erosive or atrophic forms of OLP

Exclusion Criteria:

* lichenoid lesions
* Presence of systemic conditions
* Smoking
* Known hypersensitivity or severe adverse effects to the treatment drugs or to any ingredient of their preparation
* Pregnancy or breast-feeding
* History of previous treatments potentially effective on OLP in last 3 months
* Loss of pliability or flexibility in the tissues involved by the oral lesions of lichen planus

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Clinical score | change from Baseline at 12 weeks
  "0" represented no lesion/normal mucosa; "1" mild white striae/no erythematous area, "2"white striae with atrophic area less than 1 cm², "3" white striae with atrophic area more than 1 cm², "4" white striae with erosive area less than 1 cm², and "5" white striae with erosive area more than 1 cm²

SECONDARY OUTCOMES:
IKK-alpha | change from baseline at 8 weeks
  Inhibitor kappa kinase alpha immunopositive cells count in immunostained section

OTHER OUTCOMES:
VAS | change from Baseline at 12 weeks
  Patients ranked the severity of pain on 100-mm visual analog scale
TUA | change from Baseline at 12 weeks
  Surface area of ulcer in marker lesion in mm2
TAA | change from Baseline at 12 weeks
  Surface area of atrophied red area in marker lesion in mm2
IL-8 | change from baseline at 8 weeks
  Mean area fraction of immunopositive IL-8 in section

CONTACTS AND LOCATIONS:
Overall Officials: Hala A. Abo el ela, Professor, Study Director — Faculty of dentistry- Ain shams University

IPD SHARING:
Plan to Share IPD: Undecided